CLINICAL TRIAL: NCT02585310
Title: Packed Red Blood Cell Transfusion in Elective Coronary Artery Bypass Graft Surgery in A University Hospital
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Sirilak Suksompong, Associate Professor, Mahidol University
Other Study IDs: SI1
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: PRBC Transfusion; CABGs
Keywords: PRBC transfusion; CABGs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Packed red blood cell transfusion — Record number of PRBC transfusion during perioperative period.

SUMMARY:
In Siriraj Hospital, blood consumption in Cardiac surgery is high (units per patient) and frequent (number of patients receiving blood). The incidence of side effects are unknown, as is the exact amount of blood used/provided for patients with elective CABGs.

The primary objective of this study was to demonstrate the incidence of packed red blood cell (PRBC) transfusion in elective CABGs.

DETAILED DESCRIPTION:
Three hundred patients undergoing isolated, first time CABGs during November 2011-September 2013 were prospective enrolled in this observational study. Patients' preoperative variables and postoperative outcomes, as well as perioperative transfusion characteristics were recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing first-time isolated elective coronary artery bypass graft surgery

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing CABGs
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
incidence of PRBC transfusion in elective CABG surgery | 14 days

SECONDARY OUTCOMES:
risk factors of PRBC transfusion in elective CABG surgery | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Sirilak Suksompong, MD, Principal Investigator — Mahidol University